CLINICAL TRIAL: NCT02924376
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy and Safety of Pemigatinib in Subjects With Advanced/Metastatic or Surgically Unresectable Cholangiocarcinoma Including FGFR2 Translocations Who Failed Previous Therapy - (FIGHT-202)
Brief Title: Efficacy and Safety of Pemigatinib in Subjects With Advanced/Metastatic or Surgically Unresectable Cholangiocarcinoma Who Failed Previous Therapy - (FIGHT-202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 54828-202; 2016-002422-36 (EudraCT Number)
Expanded Access: NCT03906357 (No longer available)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2023-02-23 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; fibroblast growth factor (FGF); fibroblast growth factor receptor (FGFR); FGF/FGFR alterations
MeSH Terms: conditions — Cholangiocarcinoma; Acrocephalosyndactylia | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (3):
- Cohort A Pemigatinib (Experimental): Pemigatinib in subjects with FGFR2 translocation with a documented fusion partner in central laboratory report
  Interventions: Drug: Pemigatinib
- Cohort B Pemigatinib (Experimental): Pemigatinibin subjects with other FGF/FGFR alterations
  Interventions: Drug: Pemigatinib
- Cohort C Pemigatinib (Experimental): Pemigatinib in subjects negative for FGF/FGFR alteration
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinibonce a day by mouth for 2 consecutive weeks and 1 week off therapy
  Other Names: INCB054828

SUMMARY:
The purpose of this study is evaluate the efficacy of pemigatinib in subjects with advanced/metastatic or surgically unresectable cholangiocarcinoma with FGFR2 translocation who have failed at least 1 previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cholangiocarcinoma.
* Radiographically measurable or evaluable disease per RECIST v1.1.
* Tumor assessment for FGF/FGFR gene alteration status.
* Documented disease progression after at least 1 line of prior systemic therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Life expectancy ≥ 12 weeks.

Exclusion Criteria:

* Prior receipt of a selective FGFR inhibitor.
* History of and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcifications.
* Current evidence of clinically significant corneal or retinal disorder confirmed by ophthalmologic examination.
* Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives, whichever is shorter, before the first dose of study drug. Topical ketoconazole will be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Féliz Vinas, MD, Study Director — Incyte Corporation
Locations (120):
- United States (49):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Orange, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - New Haven, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami Beach, Florida
  - Chicago, Illinois
  - Evanston, Illinois
  - Fort Wayne, Indiana
  - Sioux City, Iowa
  - Westwood, Kansas
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Rochester, Minnesota
  - Woodbury, Minnesota
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Morristown, New Jersey
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Goldsboro, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sioux Falls, South Dakota
  - Arlington, Texas
  - Dallas, Texas
  - Grapevine, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Tyler, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Fairfax, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Belgium (4):
  - Brussels
  - Ghent
  - Kortrijk
  - Leuven
- France (6):
  - Montpellier, Herault
  - Villejuif, Herault
  - Avignon
  - Clichy
  - Paris
  - Toulouse
- Germany (8):
  - Berlin
  - Bonn
  - Dresden
  - Hanover
  - Homburg
  - Leipzig
  - Mainz
  - Tübingen
- Israel (4):
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (14):
  - Bari, Castellana Grotte
  - San Giovanni Rotondo, Foggia
  - Bergamo
  - Bologna
  - Candiolo
  - Catania
  - Faenza
  - Lecce
  - Meldola
  - Milan
  - Napoli
  - Rimini
  - Siena
  - Verona
- Japan (11):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Yokohama, Kanagawa
  - Kyoto, Kyoto
  - Osaka, Osaka
  - Osakasayama-shi, Osaka
  - Kitaadachi, Saitama
  - Sunto, Shizuoka
  - Kōtoku, Tokyo-To
  - Shinjuku-ku, Tokyo-To
- South Korea (3):
  - Goyang-si
  - Seongnam-si
  - Seoul
- Spain (4):
  - Pamplona, Navarre
  - Barcelona
  - Girona
  - Madrid
- Taiwan (3):
  - Taichung
  - Tainan
  - Taipei
- Thailand (5):
  - Chiang Mai, Muang
  - Khon Kaen, Muang
  - Udon Thani, Muang
  - Bangkok, Patumwan
  - Bangkoknoi
- United Kingdom (9):
  - Cambridge, Cambridgeshire
  - Bournemouth, Dorset
  - Aberdeen, Grampian Region
  - London, Greater London
  - Cardiff
  - Glasgow
  - Manchester
  - Metropolitan Borough of Wirral
  - Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- [Derived] Patel TH, Marcus L, Horiba MN, Donoghue M, Chatterjee S, Mishra-Kalyani PS, Schuck RN, Li Y, Zhang X, Fourie Zirkelbach J, Charlab R, Liu J, Yang Y, Lemery SJ, Pazdur R, Theoret MR, Fashoyin-Aje LA. FDA Approval Summary: Pemigatinib for Previously Treated, Unresectable Locally Advanced or Metastatic Cholangiocarcinoma with FGFR2 Fusion or Other Rearrangement. Clin Cancer Res. 2023 Mar 1;29(5):838-842. doi: 10.1158/1078-0432.CCR-22-2036. PMID 36206041
- [Derived] Bibeau K, Feliz L, Lihou CF, Ren H, Abou-Alfa GK. Progression-Free Survival in Patients With Cholangiocarcinoma With or Without FGF/FGFR Alterations: A FIGHT-202 Post Hoc Analysis of Prior Systemic Therapy Response. JCO Precis Oncol. 2022 Apr;6:e2100414. doi: 10.1200/PO.21.00414. PMID 35544727
- [Derived] Abou-Alfa GK, Sahai V, Hollebecque A, Vaccaro G, Melisi D, Al-Rajabi R, Paulson AS, Borad MJ, Gallinson D, Murphy AG, Oh DY, Dotan E, Catenacci DV, Van Cutsem E, Ji T, Lihou CF, Zhen H, Feliz L, Vogel A. Pemigatinib for previously treated, locally advanced or metastatic cholangiocarcinoma: a multicentre, open-label, phase 2 study. Lancet Oncol. 2020 May;21(5):671-684. doi: 10.1016/S1470-2045(20)30109-1. Epub 2020 Mar 20. PMID 32203698

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled participants at 68 study sites in the United States, South Korea, United Kingdom, France, Italy, Thailand, Germany, Belgium, Israel, Spain, Japan, and Taiwan.
Groups:
- Cohort A: FGFR2 Rearrangements or Fusions: Participants with fibroblast growth factor (FGF) receptor 2 (FGFR2) rearrangements or fusions self-administered oral pemigatinib at a starting dose of 13.5 milligrams (mg) once daily (QD) on a 2-weeks-on therapy/1-week-off schedule in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
- Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions: Participants with all other FGF/FGFR alterations self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a 2-weeks-on therapy/1-week-off schedule in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
- Cohort C: Negative for FGF/FGFR Alterations: Participants with no FGF/FGFR alterations self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a 2-weeks-on therapy/1-week-off schedule in 21-day cycles (United States only). Pemigatinib was administered until documented disease progression or unacceptable toxicity.
- Other: Participants with an FGF/FGFR status for whom the local laboratory FGF/FGFR results could not be confirmed centrally self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a 2-weeks-on therapy/1-week-off schedule in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Started | 108 | 20 | 17 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 108 | 20 | 17 | 2
Not completed — Progressive Disease | 4 | 0 | 1 | 0
Not completed — Death | 73 | 18 | 15 | 2
Not completed — Lost to Follow-up | 3 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 19 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 1 | 0
Not completed — Rolled Over to Another Study | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other | Total
Number analyzed (Participants) | 108 | 20 | 17 | 2 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.00) | 61.9 (10.99) | 65.6 (7.12) | 41.0 (14.14) | 57.1 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 11 | 7 | 1 | 85
  Male | 42 | 9 | 10 | 1 | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 79 | 9 | 14 | 2 | 104
  Black or African American | 7 | 0 | 1 | 0 | 8
  Asian | 12 | 11 | 0 | 0 | 23
  American-Indian/Alaska Native | 0 | 0 | 1 | 0 | 1
  Captured as "Other" | 4 | 0 | 1 | 0 | 5
  Missing | 6 | 0 | 0 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 4 | 0 | 6
  Not Hispanic or Latino | 88 | 18 | 13 | 2 | 121
  Not Reported | 15 | 0 | 0 | 0 | 15
  Unknown | 1 | 0 | 0 | 0 | 1
  Captured as "Other" | 2 | 2 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in Participants With FGFR2 Rearrangements or Fusions
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) at any post-Baseline visit prior to first progressive disease (PD), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. ORR was based on central genomics laboratory results. Response was based on review of scans by an independent centralized radiological review committee.
Time Frame: up to 1527 days
Population: Efficacy Evaluable Population (EEP): all participants who received ≥1 dose of pemigatinib and had a known FGF/FGFR alteration or, in the United States, were negative for FGF/FGFR alterations based on central genomics laboratory results. Two participants were assigned to a group labeled "Other" and were excluded from the EEP because the local laboratory FGF/FGFR results could not be confirmed centrally. Confidence intervals were calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 108 | 0 | 0 | 0
percentage of participants | 37.0 [27.94 to 46.86] |  |  |

2. Secondary Outcome: ORR in Participants FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions
Description: ORR was defined as the percentage of participants with a best overall response of CR or PR at any post-Baseline visit prior to first PD, per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. ORR was based on central genomics laboratory results. Response was based on review of scans by an independent centralized radiological review committee.
Time Frame: up to 424 days
Population: Efficacy Evaluable Population. Two participants were assigned to a group labeled "Other" and were excluded from the EEP because the local laboratory FGF/FGFR results could not be confirmed centrally. Confidence intervals were calculated based on the exact method for binomial distribution.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 0 | 20 | 0 | 0
percentage of participants |  | 0.0 [0.0 to 16.84] |  |

3. Secondary Outcome: ORR in All Participants With FGF/FGFR Alterations
Description: as for outcome 2
Time Frame: up to 1527 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A + Cohort B: Participants with FGFR2 rearrangements or fusions (Cohort A) or with all other FGF/FGFR alterations (Cohort B) self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a 2-weeks-on therapy/1-week-off schedule in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other | Cohort A + Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 128
percentage of participants |  |  |  |  | 31.3 [23.35 to 40.04]

4. Secondary Outcome: ORR in Participants Negative for FGF/FGFR Alterations
Description: as for outcome 2
Time Frame: up to 143 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 0 | 0 | 17 | 0
percentage of participants |  |  | 0.0 [0.0 to 19.51] |

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the length of time from the first dose of study drug (Day 1) to the earlier of death or disease progression by RECIST v1.1, as assessed by the independent centralized radiological review committee.
Time Frame: up to 50.17 months
Population: Efficacy Evaluable Population. Two participants were assigned to a group labeled "Other" and were excluded from the EEP because the local laboratory FGF/FGFR results could not be confirmed centrally. The 95% confidence intervals were calculated using the Brookmeyer and Crowley's method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 108 | 20 | 17 | 0
months | 7.03 [6.08 to 10.48] | 2.10 [1.18 to 4.86] | 1.51 [1.38 to 1.84] |

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first overall response contributing to an objective response (CR or PR) as assessed by an independent centralized radiological review committee to the earlier of death or first overall response of PD occurring after the first overall response contributing to the objective response. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion.
Time Frame: up to 47.11 months
Population: Efficacy Evaluable Population. Two participants were assigned to a group labeled "Other" and were excluded from the EEP because the local laboratory FGF/FGFR results could not be confirmed centrally. The 95% confidence intervals were calculated using the Brookmeyer and Crowley's method. Only participants with a CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 40 | 0 | 0 | 0
months | 9.13 [6.01 to 14.49] |  |  |

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants with an overall response of CR, PR, or stable disease (SD), per RECIST v1.1. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 1527 days
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 108 | 20 | 17 | 0
percentage of participants | 82.4 [73.9 to 89.1] | 40.0 [19.1 to 63.9] | 17.6 [3.8 to 43.4] |

8. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the length of time from the first dose of study drug (Day 1) until the date of death due to any cause.
Time Frame: up to 51.32 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 108 | 20 | 17 | 0
months | 17.48 [14.36 to 22.93] | 6.70 [2.10 to 10.55] | 3.98 [1.97 to 4.60] |

9. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any adverse event either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and within 30 days of the last dose of study drug.
Time Frame: up to 1584 days
Population: Safety Population: all enrolled participants who received at least 1 dose of pemigatinib
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other
Number analyzed (Participants) | 108 | 20 | 17 | 2
Participants | 108 | 20 | 17 | 2

10. Secondary Outcome: First-order Absorption Rate Constant (ka) of Pemigatinib
Description: First-order absorption rate constant is defined as the rate at which a drug enters into the system.
Time Frame: Predose; 1-2 hours post-dose; 4-12 hours post-dose
Population: Pharmacokinetic (PK) Population: all participants contributing at least one sample for PK analysis
Measure: Mean (Standard Deviation); unit: 1/hour
Groups:
- All Cohorts: Participants with FGFR2 rearrangements or fusions (Cohort A), participants with all other FGF/FGFR alterations (Cohort B), participants with no FGF/FGFR alterations (Cohort C; United States only), and participants with an FGF/FGFR status for whom the local laboratory FGF/FGFR results could not be confirmed centrally (Other) self-administered oral pemigatinib at a starting dose of 13.5 mg QD on a 2-weeks-on therapy/1-week-off schedule in 21-day cycles. Pemigatinib was administered until documented disease progression or unacceptable toxicity.
Arm/Group | All Cohorts
Number analyzed (Participants) | 136
1/hour | 1.29 (0.827)

11. Secondary Outcome: CL/F of Pemigatinib
Description: CL/F is defined as apparent oral clearance.
Time Frame: Predose; 1-2 hours post-dose; 4-12 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | All Cohorts
Number analyzed (Participants) | 136
Liters/hour | 12.2 (5.28)

12. Secondary Outcome: Vc/F of Pemigatinib
Description: Vc/F is defined as the apparent volume of distribution for the central compartment of pemigatinib.
Time Frame: Predose; 1-2 hours post-dose; 4-12 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | All Cohorts
Number analyzed (Participants) | 136
Liters | 144 (55.7)

13. Secondary Outcome: Vp/F of Pemigatinib
Description: Vp/F is defined as the apparent volume of distribution for the tissue (peripheral) compartment.
Time Frame: Predose; 1-2 hours post-dose; 4-12 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | All Cohorts
Number analyzed (Participants) | 136
Liters | 85.6 (30.5)

ADVERSE EVENTS:
Time Frame: up to 1584 days
Description: Treatment-emergent adverse events, defined as adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last dose of study drug, have been reported.
Groups:
- Total: Total
Arm/Group | Cohort A: FGFR2 Rearrangements or Fusions | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions | Cohort C: Negative for FGF/FGFR Alterations | Other | Total
All-Cause Mortality (participants affected / at risk) | 76/108 | 18/20 | 15/17 | 2/2 | 111/147
Serious Adverse Events (participants affected / at risk) | 46/108 | 10/20 | 12/17 | 0/2 | 68/147
Other Adverse Events (participants affected / at risk) | 108/108 | 20/20 | 17/17 | 2/2 | 147/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: FGFR2 Rearrangements or Fusions (N=108) | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions (N=20) | Cohort C: Negative for FGF/FGFR Alterations (N=17) | Other (N=2) | Total (N=147)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 1 (1) | 2 (2) | 0 (0) | 7 (9)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Biliary obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Biliary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Biloma (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 5 (8) | 0 (0) | 1 (1) | 0 (0) | 6 (9)
Cholangitis infective (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Device leakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 5 (5)
Pneumonia (Infections and infestations) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (7) | 1 (1) | 1 (1) | 0 (0) | 7 (9)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (5) | 0 (0) | 1 (2) | 0 (0) | 3 (7)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: FGFR2 Rearrangements or Fusions (N=108) | Cohort B: FGF/FGFR Alterations Other Than FGFR2 Rearrangements or Fusions (N=20) | Cohort C: Negative for FGF/FGFR Alterations (N=17) | Other (N=2) | Total (N=147)
Abdominal distension (Gastrointestinal disorders) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 22 (39) | 3 (3) | 3 (3) | 1 (1) | 29 (46)
Abdominal pain upper (Gastrointestinal disorders) | 11 (16) | 2 (2) | 1 (1) | 0 (0) | 14 (19)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 5 (6) | 1 (1) | 2 (2) | 0 (0) | 8 (9)
Alanine aminotransferase increased (Investigations) | 12 (16) | 0 (0) | 1 (1) | 0 (0) | 13 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 64 (66) | 4 (4) | 3 (3) | 2 (2) | 73 (75)
Anaemia (Blood and lymphatic system disorders) | 16 (27) | 2 (2) | 2 (2) | 0 (0) | 20 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (52) | 5 (8) | 2 (3) | 0 (0) | 44 (63)
Ascites (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 9 (16) | 1 (3) | 2 (2) | 0 (0) | 12 (21)
Asthenia (General disorders) | 15 (34) | 4 (9) | 1 (1) | 0 (0) | 20 (44)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (34) | 1 (1) | 2 (2) | 0 (0) | 30 (37)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood 1,25-dihydroxycholecalciferol decreased (Investigations) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Blood 1,25-dihydroxycholecalciferol increased (Investigations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 12 (16) | 1 (1) | 2 (2) | 0 (0) | 15 (19)
Blood bilirubin increased (Investigations) | 6 (9) | 0 (0) | 1 (1) | 0 (0) | 7 (10)
Blood chloride decreased (Investigations) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 2 (5)
Blood creatinine increased (Investigations) | 9 (12) | 2 (2) | 4 (4) | 0 (0) | 15 (18)
Blood parathyroid hormone decreased (Investigations) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 4 (6)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
C-reactive protein increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 7 (10)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Chills (General disorders) | 6 (8) | 0 (0) | 2 (2) | 0 (0) | 8 (10)
Cholangitis (Hepatobiliary disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Chorioretinal scar (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Conjunctivitis (Infections and infestations) | 7 (9) | 1 (1) | 1 (1) | 0 (0) | 9 (11)
Constipation (Gastrointestinal disorders) | 46 (68) | 5 (6) | 2 (2) | 1 (1) | 54 (77)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 0 (0) | 2 (2) | 0 (0) | 12 (14)
Cystitis (Infections and infestations) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 34 (39) | 7 (10) | 7 (8) | 1 (2) | 49 (59)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 16 (17) | 1 (2) | 3 (4) | 1 (1) | 21 (24)
Depression (Psychiatric disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 9 (9)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 58 (169) | 5 (15) | 6 (6) | 1 (1) | 70 (191)
Dizziness (Nervous system disorders) | 19 (23) | 1 (1) | 1 (1) | 0 (0) | 21 (25)
Dry eye (Eye disorders) | 38 (45) | 1 (1) | 1 (1) | 1 (1) | 41 (48)
Dry mouth (Gastrointestinal disorders) | 42 (49) | 5 (5) | 1 (1) | 2 (2) | 50 (57)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (33) | 0 (0) | 0 (0) | 2 (2) | 32 (35)
Dysgeusia (Nervous system disorders) | 45 (49) | 3 (5) | 3 (3) | 2 (2) | 53 (59)
Dyspepsia (Gastrointestinal disorders) | 14 (17) | 2 (2) | 0 (0) | 0 (0) | 16 (19)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 3 (3) | 3 (3) | 0 (0) | 16 (18)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Dysuria (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 1 (1) | 0 (0) | 0 (0) | 20 (25)
Erythema (Skin and subcutaneous tissue disorders) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Eye discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 8 (13) | 0 (0) | 1 (1) | 0 (0) | 9 (14)
Fatigue (General disorders) | 50 (60) | 5 (6) | 9 (9) | 0 (0) | 64 (75)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 7 (7)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 (14) | 1 (1) | 2 (2) | 0 (0) | 16 (17)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Growth of eyelashes (Eye disorders) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 20 (32) | 1 (1) | 2 (2) | 0 (0) | 23 (35)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 (9) | 2 (2) | 1 (1) | 0 (0) | 12 (12)
Hypercalcaemia (Metabolism and nutrition disorders) | 16 (18) | 4 (5) | 1 (2) | 0 (0) | 21 (25)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 60 (109) | 13 (14) | 12 (13) | 1 (1) | 86 (137)
Hypertension (Vascular disorders) | 9 (11) | 3 (4) | 0 (0) | 0 (0) | 12 (15)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3) | 1 (1) | 1 (1) | 9 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 7 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 10 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (10) | 4 (6) | 4 (6) | 0 (0) | 14 (22)
Hypophosphataemia (Metabolism and nutrition disorders) | 28 (49) | 4 (6) | 2 (2) | 0 (0) | 34 (57)
Hypotension (Vascular disorders) | 5 (9) | 2 (2) | 2 (3) | 0 (0) | 9 (14)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Insomnia (Psychiatric disorders) | 13 (13) | 2 (2) | 0 (0) | 0 (0) | 15 (15)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 7 (12) | 0 (0) | 0 (0) | 0 (0) | 7 (12)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5) | 1 (2) | 1 (1) | 0 (0) | 6 (8)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (12) | 1 (1) | 1 (1) | 0 (0) | 13 (14)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (19) | 1 (1) | 2 (2) | 0 (0) | 18 (22)
Nail discolouration (Skin and subcutaneous tissue disorders) | 12 (12) | 1 (1) | 0 (0) | 1 (1) | 14 (14)
Nail disorder (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 11 (14) | 1 (1) | 0 (0) | 0 (0) | 12 (15)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 1 (1) | 2 (2) | 0 (0) | 11 (12)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 0 (0) | 0 (0) | 0 (0) | 13 (14)
Nasopharyngitis (Infections and infestations) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Nausea (Gastrointestinal disorders) | 45 (71) | 7 (10) | 7 (7) | 1 (2) | 60 (90)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 7 (7)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 9 (10)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 5 (6)
Ocular hyperaemia (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Oedema peripheral (General disorders) | 16 (21) | 4 (4) | 6 (6) | 0 (0) | 26 (31)
Onychoclasis (Skin and subcutaneous tissue disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 9 (10)
Onycholysis (Skin and subcutaneous tissue disorders) | 10 (10) | 2 (2) | 1 (1) | 0 (0) | 13 (13)
Onychomadesis (Skin and subcutaneous tissue disorders) | 13 (14) | 1 (1) | 0 (0) | 0 (0) | 14 (15)
Oral candidiasis (Infections and infestations) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 2 (2) | 0 (0) | 0 (0) | 13 (15)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (41) | 3 (4) | 0 (0) | 0 (0) | 29 (45)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 23 (34) | 1 (2) | 0 (0) | 0 (0) | 24 (36)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Paronychia (Infections and infestations) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 10 (10)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Platelet count decreased (Investigations) | 8 (15) | 1 (1) | 0 (0) | 1 (1) | 10 (17)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Presbyopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (15) | 1 (1) | 1 (1) | 0 (0) | 15 (17)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Punctate keratitis (Eye disorders) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 10 (10)
Pyrexia (General disorders) | 11 (20) | 3 (3) | 2 (2) | 0 (0) | 16 (25)
Rash (Skin and subcutaneous tissue disorders) | 12 (14) | 0 (0) | 1 (1) | 0 (0) | 13 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 7 (7)
Skin fissures (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 46 (74) | 6 (10) | 3 (3) | 1 (1) | 56 (88)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subretinal fluid (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Taste disorder (Nervous system disorders) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Transaminases increased (Investigations) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 4 (6)
Tri-iodothyronine free increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 11 (11) | 2 (2) | 0 (0) | 0 (0) | 13 (13)
Trichomegaly (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Trichomoniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Urinary tract infection (Infections and infestations) | 21 (33) | 2 (3) | 2 (2) | 1 (1) | 26 (39)
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 10 (10) | 1 (1) | 0 (0) | 1 (1) | 12 (12)
Vitreous floaters (Eye disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 6 (7)
Vomiting (Gastrointestinal disorders) | 35 (55) | 3 (3) | 4 (5) | 0 (0) | 42 (63)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 20 (23) | 4 (4) | 1 (1) | 1 (1) | 26 (29)
Weight increased (Investigations) | 4 (7) | 1 (2) | 0 (0) | 0 (0) | 5 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT02924376/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT02924376/SAP_001.pdf